CLINICAL TRIAL: NCT01205828
Title: Phase II Study of ABT-888 and Temozolomide in Patients With Advanced Hepatocellular Carcinoma (HCC) Progressing Following Sorafenib Treatment or Intolerant to Sorafenib
Brief Title: ABT-888 and Temozolomide for Liver Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Georgetown University (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-268
Record Dates: First submitted 2010-09-18; First posted 2010-09-21 (Estimated); Results first posted 2016-04-01 (Estimated); Last update posted 2025-02-12 (Actual); Status verified 2017-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: liver cancer; hepatocellular; temozolomide; veliparib
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Temozolomide; veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Temozolomide and ABT-888 in HCC patients (Experimental): Temozolomide 150 mg/m2/day PO Days 1-5 every 28 days ABT-888 40 mg BID PO Days 1-7 every 28 days
  Interventions: Drug: Temozolomide; Drug: ABT-888

INTERVENTIONS:
Drug: Temozolomide — Temozolomide 150 mg/m2/day PO Days 1-5 every 28 days
  Other Names: Temodar
Drug: ABT-888 — ABT-888 40 mg BID PO Days 1-7 every 28 days
  Other Names: Veliparib

SUMMARY:
This study is for people with liver cancer (also called hepatocellular carcinoma, or HCC in abbreviation).

The purpose of this study is to test the efficacy (effectiveness) of a new combination of drugs, ABT-888 and temozolomide for patients with liver cancer. Temozolomide acts by damaging deoxyribonucleic acid (DNA) in rapidly dividing cells, in other words, cancer cells. ABT-888 inhibits an enzyme called "PARP" which helps to fix damaged DNA. By inhibiting this enzyme, ABT-888 prevents cancer cells from repairing the damage caused by the temozolomide and will hopefully increase the killing of cancer cells, and decrease the tumors in the body.

ABT-888 is an investigational or experimental anti-cancer agent that has not yet been approved by the Food and Drug Administration (FDA) for use in liver cancer.

This study will help find out what effects (good and bad) the combination of drugs, temozolomide and ABT-888, has on liver cancer.

This research is being done because it is not known if ABT-888 will increase the effectiveness of temozolomide in liver cancer.

DETAILED DESCRIPTION:
Patients with hepatocellular carcinoma seen at Lombardi Cancer Center were evaluated for the eligibility of this study.

The Georgetown Lombardi Comprehensive Cancer Center was responsible for the data and safety monitoring of this trial. As this study is an investigator initiated study Phase II study utilizing a non-FDA approved drug for which the PI held the IND it was considered a high risk study which had real-time monitoring by the PI and study team and quarterly reviews by the LCCC Data and Safety Monitoring Committee (DSMC).

ELIGIBILITY:
Inclusion Criteria:

* Pathological confirmation of HCC or noninvasive criteria following AASLD guidelines
* Measurable or evaluable disease based on RECIST criteria
* Progressive disease on sorafenib or intolerance to sorafenib
* ECOG performance status 0-2
* Child Pugh Class A or B
* Adequate hepatic, bone marrow, and renal function

Exclusion Criteria:

* Prior ABT-888 or other PARP inhibitor treatment
* Anticipation of need for major surgery during the study
* Any of the following within 6 months before enrollment: myocardial infarction, severe/unstable angina, congestive heart failure, or severe pulmonary disease
* Women who are pregnant or lactating
* Women and men of child-bearing potential who are not using a reliable form of contraception
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ABT-888 and temozolomide
* Concurrent malignancy (i.e. malignancy other than hepatocellular cancer) unless 1) the subject has been curatively treated and disease free for at least 2 years or 2) the cancer was non-melanoma skin cancer or early cervical cancer.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (excluding active hepatitis B or C) or psychiatric illness/ social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aiwu R He, MD PhD, Principal Investigator — Georgetown University
Locations (1):
- Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Gabrielson A, Tesfaye AA, Marshall JL, Pishvaian MJ, Smaglo B, Jha R, Dorsch-Vogel K, Wang H, He AR. Phase II study of temozolomide and veliparib combination therapy for sorafenib-refractory advanced hepatocellular carcinoma. Cancer Chemother Pharmacol. 2015 Nov;76(5):1073-9. doi: 10.1007/s00280-015-2852-2. Epub 2015 Oct 8. PMID 26449224

RESULTS

PARTICIPANT FLOW:
Groups:
- ABT-888 and Temozolomide: ABT-888 40 mg daily day 1-7/28 and temozolomide 150 mg/m2/day day 1-5/28
Period: Overall Study
Arm/Group | ABT-888 and Temozolomide
Started | 16
Completed | 16 (Completed the first stage of the study, terminated as pre-planned due to lack of efficacy)
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Temozolomide + ABT-888: Temozolomide and ABT-888
  temozolomide + ABT-888: Temozolomide 150 mg/m2/day PO Days 1-5 every 28 days ABT-888 40 mg BID PO Days 1-7 every 28 days
  Patents with stable disease or continued response to therapy will be treated and followed for a total of 6 cycles (6 months).
Arm/Group | Temozolomide + ABT-888
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 61 [40 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 4
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate
Description: complete response at any time + partial response at any time + stable disease after 8 weeks of treatment based on RECIST Criteria
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | ABT-888 and Temozolomide
Number analyzed (Participants) | 16
participants | 3

2. Secondary Outcome: Overall Survival
Description: the number of months between a patient's enrollment and his/her date of death
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ABT-888 and Temozolomide
Number analyzed (Participants) | 16
months | 13.1 [1 to 32.0]

3. Secondary Outcome: Progression Free Survival
Description: The number of months between a patient's enrollment and his/her disease progression
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ABT-888 and Temozolomide
Number analyzed (Participants) | 16
months | 1.9 [1.8 to 2.0]

4. Secondary Outcome: Number of Participants Who Had Grade 3 or 4 Adverse Events
Description: Record of all toxicities graded according to the NCI CTCAE version 3.0
Time Frame: 6 months
Population: grade 3 or 4 adverse events
Measure: Number; unit: participants
Arm/Group | ABT-888 and Temozolomide
Number analyzed (Participants) | 16
participants | 5

5. Secondary Outcome: Biomarker Analysis
Description: To evaluate biological correlation with response to ABT-888 and temozolomide, including evaluation of loss of heterozygosity (LOH) of 13q, decreased expression of or mutations in BRCA-1 or -2, and a select assortment of DNA repair genes.
Time Frame: 6 months
Population: Since the treatment showed no significant efficacy against HCC, therefore study of biomarker that predict responsiveness of the treatment was not carried out.
Arm/Group | Temozolomide and ABT-888 in HCC Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Temozolomide + ABT-888
Serious Adverse Events (participants affected / at risk) | 6/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide + ABT-888 (N=16)
nausea, vomit (Gastrointestinal disorders) | 3 (4)
fatigue (General disorders) | 1 (1)
bleeding (Gastrointestinal disorders) | 1 (1) — rupture of the primary tumor
multiorgan failure (Renal and urinary disorders) | 1 (1) — hepato-renal syndrome from large quantity paracentesis
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide + ABT-888 (N=16)
fatigue (General disorders) | 7 (7)
platelet count decrease (Blood and lymphatic system disorders) | 6 (6)
low neutrophil (Blood and lymphatic system disorders) | 4 (4)
low lymphocyte (Blood and lymphatic system disorders) | 4 (4)
nausea, vomit (Gastrointestinal disorders) | 4 (4)
diarrhea (Gastrointestinal disorders) | 2 (2)
constipation (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days